CLINICAL TRIAL: NCT06316115
Title: In Patıents Wıth Dıabetıc Foot Ulcer, Effect On Paın And Anxıety Of Stress Ball Use Durıng Sharp Debrıdement
Brief Title: Effect On Paın And Anxıety Of Stress Ball Use Durıng Sharp Debrıdement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Fatma Aslan, Lecturer, Harran University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HRRU-KMY-FA-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: diabetic food ulcer; stress ball; pain; anxciety
MeSH Terms: conditions — Diabetic Foot; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wound debridement of patients with diabetic foot ulcers (No Intervention): No Intervention: The patient's pain and anxiety will be evaluated by a nurse independent of the research before and during the debridement procedure, without any intervention to the patients
- Patients with diabetic foot ulcers using stress balls during wound debridement (Experimental): Intervention Group: Patients in this group participating in the study will be given a stress ball and asked to use it before the debridement procedure, and each patient will be debrided by the same person throughout the procedure. The patient's pain and anxiety will be evaluated by a nurse independent of the research before and after the debridement procedure.
  Interventions: Other: In Patıents Wıth Dıabetıc Foot Ulcer, Effect On Paın And Anxıety Of Stress Ball Use Durıng Sharp Debrıdement

INTERVENTIONS:
Other: In Patıents Wıth Dıabetıc Foot Ulcer, Effect On Paın And Anxıety Of Stress Ball Use Durıng Sharp Debrıdement — Patients in this group participating in the study will be given a stress ball and asked to use it before the debridement procedure, and each patient will be debrided by the same person throughout the procedure. The patient's pain and anxiety will be evaluated by a nurse independent of the research before and after the debridement procedure.
  Arms: Patients with diabetic foot ulcers using stress balls during wound debridement

SUMMARY:
Diabetic foot ulcer; It is a disease used to describe a series of lower extremity complications that may occur together with infection, ulceration or gangrene in individuals with diabetes and is coded as S91.3 and S91.8 in the International Classification of Diseases (ICD). Sharp debridement, one of the treatments for diabetic foot ulcers, is a short-term application performed with a sharp scalpel or scissors at the patient's bed or in outpatient clinic conditions. It should be performed by a skilled clinician with wound training. To our knowledge, no study has been found in the literature regarding the use of a stress ball as an intervention to prevent pain and anxiety during sharp debridement. In line with this information, this study will examine the effect of stress ball use on the pain and anxiety levels of patients with diabetic foot ulcers during wound debridement.

DETAILED DESCRIPTION:
The annual number of patients hospitalized with diabetic foot ulcer treatment is 543, and the sample calculation of the study was determined using the G*Power program. Since there was no previous study conducted in the same study group, a study examining the effect of stress ball on pain in invasive procedures was taken as reference in the calculation of the sample. In this study, it was predicted that the difference between pain intensities would be evaluated with a t test, and the effect value was predicted to be 0.70 with a 95% confidence interval and 80% power, and it was calculated that 34 participants would be sufficient for the sample. Considering possible losses from the study (hospitalization, death, changing treatment center, etc.), a total of 76 patients, 38 in each group, were aimed to be included in the study.

As a data collection tool; Introductory Information Form, Meggit-Wagner Classification, Visual Comparison Scale and State Anxiety Scale (STAI) will be used.

Intervention Group: Patients in this group participating in the study will be given a stress ball and asked to use it before the debridement procedure, and each patient will be debrided by the same person throughout the procedure. The patient's pain and anxiety will be evaluated by a nurse independent of the research before and after the debridement procedure.

Control Group: The patient's pain and anxiety will be evaluated by a nurse independent of the research before and during the debridement procedure, without any intervention to the patients.

Stress ball use: Before starting the study, the researchers explained to the patients theoretically how to use the stress ball and demonstrated it practically. Then, the patient was asked to use the ball and it was confirmed whether he was using it correctly. Patients will be asked to count to three, squeeze the ball once and then relax it, inhale each time they squeeze the ball, and exhale when they relax it. The stress ball used is made of medium hardness and high quality silicone. The balls will be provided by the researchers and given to the patients. Patients will use the stress ball throughout the debridement procedure and will continue to use it until the procedure is completed. Statistical significance level will be accepted as p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Being an inpatient in the endocrinology clinic,
* Volunteer,
* No communication problems (No hearing, understanding and speaking problems),
* Being a patient diagnosed with diabetic foot ulcer,
* The physician decided to apply sharp debridement,
* Having pain according to the Visual Comparison Scale before the sharp debridement procedure,
* Not having a health problem with the hand that would prevent him from using the ball

Exclusion Criteria:

* No pain according to the Visual Comparison Scale,
* Before performing sharp debridement, an intervention decision was taken to reduce pain (local anesthesia).
* administered, nerve blockade, opioid analgesics, etc.) excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-03-10 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | at enrollment
  Introductory information formula section by examining studies conducted with products diagnosed with diabetic foot ulcers. Promotional information regime; People's birth year, education level, employment status, income level, place of residence, year of diabetes diagnosis, etc. A total of 13 questions will be asked about.

SECONDARY OUTCOMES:
Meggit-Wagner classification of diabetic foot | baseline
  This classification system, which is based on the depth of the wound and graded in six categories from stage 0 to stage 5 according to the presence of osteomyelitis and gangrene, is evaluated with observational findings, excluding the depth of injuries. There are no limits of ischemia and cryptocurrencies and there is no presence of neuropathy. However, the positive effects of considering this in the improvement process of diabetic foot killing are known. The classification of the wound will be evaluated by a specialist physician and recorded by a certificate independent of the research. Higher scores mean a worse outcome for diabetic food ulcer.

OTHER OUTCOMES:
Visual Comparison Scale | immediately before and after the procedure
  On a scale from 0 to 10, 0 = no pain and 10 = unbearable pain. The severity of the patient's pain will be recorded before and during debridement (when the patient feels the pain decrease or increase) by a nurse independent of the study
State Anxiety scale (STAI) | immediately before and after the procedure
  Anxiety level is scored as "(1) not at all, (2) a little, (3) a lot and (4) completely" in STAI-I. Items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18 in the inventory are positive for 40 (increasing the total anxiety score), 1, 2, 5, 8, 10, 11, 15, 16, Negative scoring (reducing the total anxiety score) is given for items 19 and 20. The total score for reverse expressions is subtracted from the total score obtained for direct expressions. In scoring, a score between 1 (or -1) and 4 (or -4) is expected for each item, depending on the positive or negative feature of the item, and 50 is added to the total score to be obtained. The highest score is 80, the lowest score is 20. The higher the total anxiety score, the higher the person's anxiety level is interpreted. Before and during debridement, the State Anxiety Scale will be evaluated and recorded by a nurse independent of the research.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma ASLAN, Principal Investigator — Harran Universty
Locations (1):
- Harran Universitesi, Sanliurfa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bagcivan G, Ozen N, Bayrak D, Cinar FI. Does Being A Cancer Patient or Family Caregiver of A Cancer Patient Affect Stem Cell Donation Awareness? Asia Pac J Oncol Nurs. 2019 Jul 3;7(1):36-43. doi: 10.4103/apjon.apjon_22_19. eCollection 2020 Jan-Mar. PMID 31879682
- [Result] Ozen N, Berse S, Tosun B. Effects of using a stress ball on anxiety and depression in patients undergoing hemodialysis: A prospective, balanced, single-blind, crossover study. Hemodial Int. 2023 Oct;27(4):411-418. doi: 10.1111/hdi.13102. Epub 2023 Jun 15. PMID 37318078
- [Derived] Aslan F, Tosun B, Altinok Ersoy N, Ozen N. The effect of a stress ball on pain and anxiety during sharp debridement in patients with diabetic foot ulcers: A randomized controlled, single-blind study. J Tissue Viability. 2025 May;34(2):100861. doi: 10.1016/j.jtv.2025.100861. Epub 2025 Jan 26. PMID 39892227